CLINICAL TRIAL: NCT00273039
Title: A Randomized, Double-Blind, Parallel Group, Placebo-Controlled, Forced Dose Titration Study Evaluating the Efficacy and Safety of GW679769 and Paroxetine in Subjects With Social Anxiety Disorder
Brief Title: A Study Of A New Medicine (GW679769) For The Treatment Of Social Anxiety Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKF100110
Record Dates: First submitted 2006-01-05; First posted 2006-01-09 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Social Anxiety Disorder; Anxiety Disorders
Keywords: Social Anxiety Disorder; Anxiety; Psychiatry
MeSH Terms: conditions — Phobia, Social; Anxiety Disorders | interventions — Paroxetine

INTERVENTIONS:
Drug: paroxetine

SUMMARY:
The purpose of this study is to test the safety and efficacy of GW679769 and paroxetine in subjects with Social Anxiety Disorder

ELIGIBILITY:
Inclusion Criteria:

* Patients with Generalized Social Anxiety Disorder as the primary diagnosis.
* If female, must commit to consistent and correct use of an acceptable method of birth control.

Exclusion Criteria:

* Patients with any other psychiatric disorder as a primary diagnosis or within 6 months prior to screening.
* Patients with Body Dysmophic Disorder, Schizophrenia, Schizoaffective Disorder, or a Bipolar Disorder.
* Patients who pose a current suicidal or homicidal risk or have made a suicide attempt within the past 6 months or have ever been homicidal.
* Patients who have a positive urine test at screen for illegal drug use and/or a history of substance abuse or dependence (alcohol or drugs) within the past 12 months.
* Patients with an unstable medical disorder.
* Female patients who are pregnant, lactating, or planning to become pregnant during a specified time during the study.
* Patients who are taking other psychoactive medications.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 242 (Actual)
Dates: Start 2005-08; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure will be the change from baseline in the Liebowitz Social Anxiety Scale (LSAS)

SECONDARY OUTCOMES:
Secondary outcome measures include the change from baseline in the following scales: the Clinical Global Impression-Global Improvement, the Clinical Global Impression -Severity of Illness, and the Sheehan Disability Scale.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (26):
- United States (13):
  - GSK Investigational Site, Beverly Hills, California
  - GSK Investigational Site, Burbank, California
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, North Miami, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Smyrna, Georgia
  - GSK Investigational Site, Oakbrook Terrace, Illinois
  - GSK Investigational Site, Rockville, Maryland
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Lake Jackson, Texas
- Argentina (4):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, La Plata/Buenos Aires, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Buenos Aires
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Kelowna, British Columbia
  - GSK Investigational Site, Miramichi, New Brunswick
- Chile (2):
  - GSK Investigational Site, Providencia / Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Costa Rica (2):
  - GSK Investigational Site, San José, Provincia de San José
  - GSK Investigational Site, San José
- Mexico (2):
  - GSK Investigational Site, Monterrey, Nuevo León
  - GSK Investigational Site, Mexico City

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: NKF100110 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKF100110 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKF100110 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKF100110 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKF100110 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKF100110 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKF100110 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register